CLINICAL TRIAL: NCT07264855
Title: Comparison of the Effects of M-TAPA Versus the Combination of M-TAPA and EXOP Blocks on Postoperative Pain in Laparoscopic Gynecologic Surgeries
Brief Title: M-TAPA vs. Combined M-TAPA + EXOP for Postoperative Pain in Laparoscopic Gynecologic Surgery
Status: Recruiting | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Güneş Özlem Yıldız, Associate Professor, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2025/312
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain; Laparoscopic Gynecologic Surgery
Keywords: M-TAPA block; External Oblique Plane Block (EXOP); Postoperative pain; Laparoscopic gynecologic surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group M: Participants who received a bilateral M-TAPA block performed pre-extubation as part of routine anesthesia practice.
  Interventions: Procedure: Modified Thoracoabdominal Nerve Block Through Perichondrial Approach
- Group E: Participants who received a combined bilateral M-TAPA block and external oblique plane (EXOP) block performed pre-extubation as part of routine anesthesia practice.
  Interventions: Procedure: Modified Thoracoabdominal Nerve Block Through Perichondrial Approach And External Oblique Muscle Plane Block

INTERVENTIONS:
Procedure: Modified Thoracoabdominal Nerve Block Through Perichondrial Approach — A bilateral modified thoracoabdominal nerve block through the perichondrial approach (M-TAPA) is performed under ultrasound guidance in the supine position prior to extubation as part of routine clinical practice. After aseptic preparation, a linear ultrasound probe is positioned at the level of the 10th rib in the sagittal plane. The needle is advanced to the fascial plane between the internal oblique and transversus abdominis muscles. Following negative aspiration and confirmation of correct plane identification with hydrodissection, 20 mL of 0.25% bupivacaine is injected bilaterally (total volume 40 mL). The procedure is performed by anesthesiologists experienced in gynecologic surgery, without researcher involvement in clinical decision-making
  Other Names: M-TAPA Block
  Groups: Group M
Procedure: Modified Thoracoabdominal Nerve Block Through Perichondrial Approach And External Oblique Muscle Plane Block — Following completion of the bilateral M-TAPA block, an external oblique muscle plane (EXOP) block is performed under ultrasound guidance as part of routine clinical practice. The ultrasound probe is positioned over the lateral abdominal wall between the costal margin and iliac crest. After negative aspiration and confirmation of correct plane identification with hydrodissection, 20 mL of 0.125% bupivacaine is injected on each side into the fascial plane superficial to the external oblique muscle (total volume 80 mL).
  Other Names: M-TAPA + EXOP Block
  Groups: Group E

SUMMARY:
Laparoscopic gynecologic surgery is less invasive than open surgery, but many patients still experience pain after the procedure. M-TAPA and EXOP are ultrasound-guided regional anesthesia techniques used to reduce abdominal pain. Previous research suggests that M-TAPA provides effective pain relief on the anterior abdominal wall, while EXOP may help reduce pain in the lateral abdominal region. This study aims to determine whether combining M-TAPA with EXOP provides better postoperative pain control than using M-TAPA alone. The study will compare pain scores during the first 24 hours after surgery, the need for rescue analgesic medication, and recovery quality using the QoR-15 questionnaire. All procedures are part of routine clinical care, and no experimental drugs or devices are used.

DETAILED DESCRIPTION:
In routine practice at our institution, anesthesia clinicians performing gynecologic laparoscopic procedures administer either modified thoracoabdominal nerve block through perichondrial approach (M-TAPA Block) alone or a combination of M-TAPA and external oblique muscle plane (EXOP) blocks, based solely on individual clinician preference. The researcher does not influence this decision. Among the eligible patients, those receiving either M-TAPA or M-TAPA + EXOP will be included and evaluated observationally. Block types other than these two will not be included.

All postoperative visits and clinical follow-ups are routinely conducted by the hospital's pain management team. The researcher does not intervene in these clinical processes and is only responsible for obtaining informed consent, recording demographic variables, documenting the type of block performed, administering the QoR-15 questionnaire, and evaluating sensory block distribution using the pinprick test.

Preoperative evaluation and necessary laboratory testing are carried out according to standard hospital practice by the attending anesthesiologist. The researcher obtains informed consent, records demographic data, and administers the preoperative QoR-15 questionnaire.

In the operating room, standard monitoring (non-invasive blood pressure, ECG, heart rate, and oxygen saturation) is applied, intravenous access is established, and crystalloid infusion is initiated. Anesthesia induction is performed using propofol, an opioid, and a neuromuscular blocking agent, followed by endotracheal intubation. General anesthesia is maintained with sevoflurane in an oxygen-air mixture. Laparoscopic surgery is performed with gradual CO₂ insufflation, maintaining intra-abdominal pressure below 12 mmHg.

For postoperative analgesia, all patients routinely receive 1 g intravenous paracetamol and 100 mg tramadol. After surgery, neuromuscular blockade is reversed and patients are transferred to the post-anesthesia care unit (PACU).

After surgery, patients are monitored in the PACU and transferred to the ward once their Aldrete score is ≥9. All patients receive 1 g intravenous paracetamol every 8 hours as per routine protocol. Postoperative pain is assessed by the pain team using the 0-10 Numeric Rating Scale (NRS).

Postoperative nausea and vomiting (PONV) are assessed and intravenous ondansetron 4 mg is administered for PONV ≥2. Patients without PONV are encouraged to mobilize early and resume oral intake. Discharge is permitted once symptoms resolve; however, all patients remain hospitalized for at least 24 hours.

As an additional study-related procedure, the researcher evaluates dermatomal spread using the pinprick test and administers the QoR-15 questionnaire at 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laparoscopic gynecologic surgery
* Age 18-90 years
* ASA physical status I-III

Exclusion Criteria:

* Contraindications to block procedures (coagulopathy, anticoagulant therapy, local infection at needle insertion site, etc.)
* Severe cardiac, renal, hepatic, hematologic, neurologic, or psychiatric disease
* Allergy to amide-type local anesthetics
* Chronic pain, narcotic or alcohol dependence
* BMI ≥ 35 kg/m²
* Pregnancy
* Refusal to participate
* Conversion from laparoscopy to laparotomy

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult female patients undergoing laparoscopic gynecologic surgery.
Study Population: Adult female patients undergoing laparoscopic gynecologic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Score (NRS) | 1, 2, 6, 12, and 24 hours after surgery
  Postoperative pain will be assessed using the Numeric Rating Scale (NRS, 0-10). Pain scores will be recorded at 1, 2, 6, 12, and 24 hours after surgery and will be compared between Group M and Group E.
  The Numeric Rating Scale ranges from 0 to 10 (0 = no pain, 10 = worst imaginable pain); higher scores indicate worse pain.

SECONDARY OUTCOMES:
Rescue Analgesic Requirement | First 24 hours after surgery
  The total amount of rescue analgesic medication (intravenous tramadol, mg) administered in the first 24 hours will be recorded. Requirements will be compared between Group M and Group E.
Quality of Recovery (QoR-15 Score) | Preoperative baseline and postoperative 24th hour
  The quality of recovery will be assessed using the validated QoR-15 questionnaire. Scores will be compared between Group M and Group E to evaluate the impact of each block technique on postoperative recovery.
  QoR-15 total score ranges from 0 to 150; higher scores indicate better quality of recovery

OTHER OUTCOMES:
Time to First Rescue Analgesic Request | First 24 hours after surgery
  The time interval (in minutes) from the end of surgery to the first request for rescue analgesia will be recorded. Rescue analgesia will consist of intravenous 100 mg tramadol administered when the patient reports an NRS pain score ≥ 4. Results will be compared between Group M and Group E.
Dermatomal Spread (Pinprick Test) | 1, 2, 6, 12, and 24 hours after surgery
  Sensory block distribution will be assessed using the pinprick test to evaluate dermatomal spread. Results will be compared between Group M and Group E.
Postoperative Nausea and Vomiting (PONV) Score | First 24 hours after surgery
  Postoperative nausea and vomiting will be assessed using a verbal descriptive scale from 0 to 4 (0 = none, 1 = mild, 2 = moderate, 3 = single vomiting episode, 4 = multiple vomiting episodes). Scores will be compared between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- SBÜ Bakırköy Dr. Sadi Konuk Eğitim ve Araştırma Hastanesi, Istanbul, Bakirkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study contains personal health information and no regulatory or ethics approval has been obtained for external data sharing.

REFERENCES:
- [Background] Liu S, Wang Z, Long X, Fleishman A, Huang X, Wu Q, Gershman B, Olumi AF. Single black men have the worst prognosis with localized prostate cancer. Can J Urol. 2022 Feb;29(1):10992-11002. PMID 35150221
- [Background] Tulgar S, Selvi O, Thomas DT, Deveci U, Ozer Z. Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) provides effective analgesia in abdominal surgery and is a choice for opioid sparing anesthesia. J Clin Anesth. 2019 Aug;55:109. doi: 10.1016/j.jclinane.2019.01.003. Epub 2019 Jan 9. No abstract available. PMID 30639940
- [Background] Atsumi C, Aikawa K, Takahashi K, Okada K, Morimoto Y. The comparison of postoperative analgesic requirements between modified thoracoabdominal nerve block through perichondrial approach versus wound infiltration analgesia in patients undergoing gynecological laparoscopic surgery: a retrospective, exploratory study. JA Clin Rep. 2023 Jun 24;9(1):39. doi: 10.1186/s40981-023-00632-w. PMID 37354282
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331